CLINICAL TRIAL: NCT02429492
Title: Electrophysiological Biomarkers of Spinal Neural Activity: Study in Healthy Subjects Matched to ALS Patient Group
Brief Title: Spinal Interneuron Excitability in ALS
Acronym: SpineBioMark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C14-21; 2014-A01240-47 (Other: Agence Nationale de la Sécurité des Médicaments)
Record Dates: First submitted 2014-12-29; First posted 2015-04-29 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2025-03

CONDITIONS: ALS
Keywords: Pathophysiology; Spinal interneurons; Electrophysiology; EMG; transcranial magnetic stimulation (TMS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALS patients (Experimental): Patients with amyotrophy lateral sclerosis (ALS)
  Interventions: Device: Electrophysiology
- Control subjetcs (Experimental): Neurologically intact subjects sex and age-matched to ALS patients
  Interventions: Device: Electrophysiology

INTERVENTIONS:
Device: Electrophysiology — EMG recordings conditioned by electrical peripheral nerve stimulation and/or transcranial magnetic stimulation
  Other Names: EMG

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is due to neurodegeneration of upper and lower motor neurons, leading to muscle atrophy, paralysis and death. However, there is growing evidence that interneurons involved in the gain regulation of spinal motoneuron (lower motor neurons) and in sensorimotor integration may participate in the pathogenesis of ALS. While sensory afferents in the peripheral nerve are traditionally thought to be unaffected at the beginning of the disease, diffusion MRI has revealed degeneration and demyelination of the posterior columns in the spinal cord of patients recently diagnosed with ALS, and there are sporadic reports of sensory involvement. Early alteration of the sensorimotor integration could participate to the degeneration of motor neurons and interneurons. The goal of the project is to further investigate sensorimotor integration at spinal level in human patients recently diagnosed with ALS, and to study whether an interneuron pathology could participate in ALS pathogenesis.

Our project has first an interest for the fundamental research aiming at increasing basic knowledge of pathophysiology of ALS, and specifically on the functional effects of the underlying neurodegenerative mechanisms. By testing the excitability of spinal interneurons in patients recently diagnosed, and by doing so for clinically uninvolved muscles, we will be able to evaluate whether an interneuron pathology could be involved in ALS. Our results will help to understand better the chain reactions in the neurodegenerative processes that dramatically evolve until the death of all motor neurons. Our project has also an interest for the development of therapeutic approaches for ALS. Indeed, our methods will help to determine specific electrophysiological biomarkers that will help to evaluate quantitatively spinal and corticospinal neural processes: their changes during the course of the disease (follow-up study), the effect of therapeutic agents and/or rehabilitation methods on their excitability, and their repercussions on motor neuron activity (evaluation of therapeutics). Lastly, our methods could be tested in other neuromuscular diseases to determine possible differences in spinal neural activity. Indeed, the motor dysfunction common to several neuromuscular diseases can make it difficult to make a definitive diagnosis. The development of specific biomarkers is crucial for an early diagnosis, and to evaluate the best treatment for the patients as rapidly as possible.

DETAILED DESCRIPTION:
Given the all-or-none properties of neuromuscular junctions, the electromyogram (EMG) reflects the activity of spinal motoneurons. These neurons are the last order neurons in all neural pathways involved in motor control. Modification of the afferent neural activity, whatever its level (spinal or supraspinal), will affect the excitability of spinal motoneurons and thus EMG activity. Combined with electrical and/or magnetic stimulation of peripheral nerve and/or cortical structures, it is possible to test indirectly the excitability of corticospinal and spinal reflex pathways involved in human motor control. One of the novelties is that we will investigate the interneurons that are activated by motor axons or afferents inputs from affected muscles (distal musculature: hand/wrist or foot/ankle muscles), which control clinically unaffected muscles (proximal musculature: elbow or knee muscles). This has a threefold interest i) functional exploration of clinically unaffected muscles that are never evaluated in ALS patients, ii) to better interpret the EMG signal and to better elucidate the pathophysiological mechanisms underlying the change in EMG activity, and iii) to determine if interneuron pathology manifests before detectable change in the motoneuron. The conditioned EMG and threshold tracking methods will be used to evaluate the excitability of spinal interneurons in ALS patients, as compared to sex and age-matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* speaking french
* signature of the written consent
* patients with ALS and no other motor neuron disease (ALS group)
* neurologically intact subjects (Control group)

Exclusion Criteria:

* pregnancy
* contraindication to TMS

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Excitability of spinal neurons | The participants will be invited to 4 sessions of EMG recordings whose duration will be of 2h30, within the month after inlcusion for ALS patients and within the year after inclusion for the healthy subjects
  Electromyogram (EMG) reflects the activity of spinal motoneurons which is controlled by several spinal interneurons. EMG recordings will be conditioned by electrical, magnetic or mechanical stimuli to activate spinal interneurons that controlled motoneurons and thus influence the EMG recordings. The resulting changes in EMG activity will be quantified by calculating the EMG surface area or the change in peak-to-peak amplitude of evoked potentials. 2 visits will be devoted to cervical interneurons controlling upper limbs and the 2 other visits, to lumbar interneurons controlling lower limbs. Surface areas and amplitude in ALS patients will be compared to controls

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Pradat, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Pitie Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
the results will be published in international peer-reviewed journals
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2018-2019

REFERENCES:
- [Background] Turner MR, Kiernan MC. Does interneuronal dysfunction contribute to neurodegeneration in amyotrophic lateral sclerosis? Amyotroph Lateral Scler. 2012 May;13(3):245-50. doi: 10.3109/17482968.2011.636050. Epub 2012 Mar 16. PMID 22424125
- [Result] Sangari S, Peyre I, Lackmy-Vallee A, Bayen E, Pradat PF, Marchand-Pauvert V. Transient increase in recurrent inhibition in amyotrophic lateral sclerosis as a putative protection from neurodegeneration. Acta Physiol (Oxf). 2022 Apr;234(4):e13758. doi: 10.1111/apha.13758. Epub 2022 Jan 23. PMID 34981890
- [Result] Marchand-Pauvert V, Peyre I, Lackmy-Vallee A, Querin G, Bede P, Lacomblez L, Debs R, Pradat PF. Absence of hyperexcitability of spinal motoneurons in patients with amyotrophic lateral sclerosis. J Physiol. 2019 Nov;597(22):5445-5467. doi: 10.1113/JP278117. Epub 2019 Oct 26. PMID 31523813
- See also: research team web site — https://www.lib.upmc.fr/?page_id=81